CLINICAL TRIAL: NCT03650127
Title: Returning Genome and Metabolome Data to FinTerveys 2017 Participants: P5.fi
Brief Title: Returning Genome and Metabolome Data to FinTerveys 2017 Participants: P5.fi FinTerveys Study
Acronym: P5
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Markus Perola (Other Government)
Collaborators: University of Helsinki (Other); Institute for Molecular Medicine (Other)
Responsible Party: Sponsor-Investigator, Markus Perola, Research Professor, Finnish Institute for Health and Welfare
Organization: Finnish Institute for Health and Welfare (Other Government)
Other Study IDs: 1474/6.00.00/2018
Record Dates: First submitted 2018-08-24; First posted 2018-08-28 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Coronary Heart Disease; Type 2 Diabetes; Deep Vein Thrombosis
Keywords: Genetic risk score; metabolic risk score; health promotion; web-based; intervention
MeSH Terms: conditions — Coronary Disease; Diabetes Mellitus, Type 2; Venous Thrombosis; Genetic Risk Score

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
P5.fi study - P4 together with a fifth 'P' and '.fi' for population health Finally Implemented in Finland - studies the value of returning genetic and metabolomic risk information in two diseases (coronary heart disease and type 2 diabetes) and one feature (venous thromboembolism). The hypothesis of the study is that 1) combining genetic and metabolic risk with traditional risk factors adds value to the personal risk assessment of these diseases, 2) such risk information can be provided to individuals using a web based user portal in an easily understandable and useful format, and 3) receiving genetic and metabolomic risk information has an effect on the health of the study participants.

The study is a continuation of FinHealth 2017 -study, which involved more than 7,000 Finns from around the country. The participants of FinHealth were invited to participate in P5.fi -study. The new research utilises information, samples, and measurements obtained in the FinHealth Study. Prospective clinical significance of selected genetic and metabolomic risk scores will be studied in 30.000 Finnish individuals. The study will analyze the genetic and metabolomic profile of the P5.fi participants and develop and test a protocol for returning them health related risk information. The impact of the intervention will by followed up by questionnaires and national health registers for five years.

ELIGIBILITY:
Inclusion Criteria:

- Only participants of FinHealth 2017 -study are eligible for the study

Exclusion Criteria:

- Participants not part of FinHealth 2017 -study are not eligible

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population of FinHealth 2017 -study represent the general population of Finland. All participants are over 18 years of age and have been selected randomly from the population registry. All FinHealth 2017 participants with DNA sample and permission for a re-contact were invited to P5.fi study.
Sampling Method: Probability Sample
Enrollment: 3449 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Coronary heart disease/Type 2 diabetes/Venous thromboembolism diagnosis | Measure is assessed after a year from the start of the study.
  Disease diagnosis observed from the national hospitalization and death registries.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Perola, MD, PhD, Principal Investigator — National Institute of Health and Welfare
Locations (1):
- National Institute of Health and Welfare, Helsinki, Uusimaa, Finland